CLINICAL TRIAL: NCT02108639
Title: An Open-label, Multiple-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a Fixed Dose Combination Formulation of DCV, ASV, and BMS-791325 in Subjects With Normal Renal Function and Subjects With Mild, Moderate, Severe, and End-stage Renal Dysfunction
Brief Title: To Assess the Effect of Renal Impairment on the Blood Levels of Daclatasvir (DCV), Asunaprevir (ASV) and BMS-791325 After Multiple Doses of a Fixed Dose Combination Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AI443-110
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-06

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — asunaprevir; 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCV 3DAA FDC + BMS-791325 (Experimental): Group A to D: DCV 3DAA FDC + BMS-791325 oral tablets on specific days
  Group E: DCV 3DAA FDC + BMS-791325 oral tablets on specific days
  Interventions: Drug: DCV 3DAA FDC; Drug: BMS-791325

INTERVENTIONS:
Drug: DCV 3DAA FDC
  Other Names: Fixed Dose Combination of Daclatasvir, Asunaprevir and BMS-791325
Drug: BMS-791325

SUMMARY:
Assess the effect of renal function on the blood levels of DCV, ASV, BMS-791325.

DETAILED DESCRIPTION:
IND Number: 79,599/101,943

Primary Purpose: Other - Phase 1 Clinical Pharmacology study to determine the effect of renal impairment on the exposure of DCV, ASV, BMS-791325 (fixed dosed combination) and BMS-791325 given in multiple doses

Fixed dose combination (FDC)

Fixed Dose Combination of Daclatasvir, Asunaprevir and BMS-791325 (DCV 3DAA FDC)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects in Group A must be in good health and have normal renal function
* Subjects in Groups B-E may have clinical, Electrocardiogram (ECG) and laboratory findings consistent with their degree of renal dysfunction
* Women of childbearing potential (WOCBP) and male participants must agree to follow the required contraceptive methods

Exclusion Criteria:

* Subjects in Group A must not have any significant acute or chronic illnesses
* Subjects in Groups B-E must not have uncontrolled or unstable cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematopoietic, and/or neurological disease within 6 months of screening
* Subjects in Groups B-E may not have evidence of rapidly deteriorating renal function, defined as a screening creatinine clearance (CLcr) which has decreased from a previous CLcr by 50% within the last 3 months
* Prior exposure to DCV, ASV or BMS-791325 within 3 months prior to study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for DCV, ASV, BMS-791325 and BMS-794712 | For Groups A-D: Day 1 to Day 10 and for Group E: Day 1 to Day 12
Area under the concentration-time curve in 1 dosing interval (AUC(TAU)) for DCV, ASV, BMS-791325 and BMS-794712 | For Groups A-D: Day 1 to Day 10 and for Group E: Day 1 to Day 12

SECONDARY OUTCOMES:
Concentration at 12 hours (C12) for (DCV, ASV, BMS-791325) and BMS-948158 | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Time of maximum observed concentration (Tmax) for (DCV, ASV, BMS-791325) and BMS-948158 | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Apparent total body clearance (CLT/F) for (DCV, ASV and BMS-791325 only) | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Trough observed plasma concentration (Ctrough) for (DCV, ASV, BMS-791325), BMS-794712 and BMS-948158 | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Cmax fraction unbound (Cmaxfu) for (DCV, ASV, BMS-791325), BMS-794712 and BMS-948158 | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
  BMS-948158 may also be analyzed
AUC(TAU) fraction unbound (AUC(TAU) fu) for (DCV, ASV, BMS-791325), BMS-794712 and BMS-948158 | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
  BMS-948158 may also be analyzed
Protein Binding for DCV, ASV, BMS-791325 and BMS-794712 | 1 and 4 hours postdose on Day 10 (all subjects) and Day 12 (Group E only)
Total amount recovered in urine (URt) for (DCV, ASV, BMS-791325) and BMS-794712 | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Total percent of administered dose recovered in urine (%URt) for (DCV, ASV, and BMS-791325 only) | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Renal clearance (CLR) for DCV, ASV, BMS-791325, and BMS-794712 | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Maximum observed concentration (Cmax) for BMS-948158 | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Area under the concentration-time curve in 1 dosing interval (AUC (TAU)) for BMS-948158 | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Safety based on occurrence of Adverse Event (AEs), Serious adverse event (SAEs) and AEs leading to discontinuation | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Safety based on abnormalities in vital sign measurements | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Safety based on findings on ECG measurements and physical examinations | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13
Safety based on Marked abnormalities in clinical laboratory test findings | For Groups A-D: Day 1 to Day 11 and for Group E: Day 1 to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Clinical Pharmacology Of Miami Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Davita Clinical Research, Minneapolis, Minnesota
  - New Orleans Center For Clinical Research - Knoxville, Knoxville, Tennessee

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx